CLINICAL TRIAL: NCT06740071
Title: The Application of Somatosensory Interactive Pelvic Floor Muscle Training for Stress Urinary Incontinence in Men Underwent Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yung NA, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFMT-RARP
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer (Post Prostatectomy)
Keywords: pelvic floor muscle training; post operative urinary incontinence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- standard pelvic floor muscle training group (Active Comparator)
  Interventions: Behavioral: standard pelvic floor muscle training
- somatosensory interactive pelvic floor muscle training group (Active Comparator)
  Interventions: Behavioral: somatosensory interactive pelvic floor muscle training
- standard pelvic floor muscle training combined with pelvic floor magnetic stimulation therapy group (Experimental)
  Interventions: Behavioral: somatosensory interactive pelvic floor muscle training; Procedure: pelvic floor magnetic stimulation therapy

INTERVENTIONS:
Behavioral: somatosensory interactive pelvic floor muscle training — synchronized PFMT guidance through a combination of audio and video
  Arms: somatosensory interactive pelvic floor muscle training group; standard pelvic floor muscle training combined with pelvic floor magnetic stimulation therapy group
Procedure: pelvic floor magnetic stimulation therapy — stimulation frequency was set at 10 Hz, with stimulation administered in cycles of 5 seconds on followed by 5 seconds off. Each treatment session lasted 20 minutes, conducted twice a week, for a total of 10-12 sessions
  Arms: standard pelvic floor muscle training combined with pelvic floor magnetic stimulation therapy group
Behavioral: standard pelvic floor muscle training — traditional verbal instructions and paper-based educational materials of PFMT are given to participants.
  All patients would receive PFMT under the guidance of digital rectal examination by nurses, and their pelvic floor muscle function was graded according to the Oxford Grading System (grades 0-5), ensuring the correctness of subsequent PFMT.
  Arms: standard pelvic floor muscle training group

SUMMARY:
The study aims to compare the efficacy of different pelvic floor muscle training (PFMT) modes on improving urinary incontinence (UI) recovery in prostate cancer (PCa) patients after radical prostatectomy (RP). The methods being compared include standard PFMT (S-PFMT) , a somatosensory interactive PFMT (SI-PFMT, an enhanced PFMT) , and a standard PFMT combined with pelvic floor muscle magnetic stimulation (S-PFMT+MS). Eligible participants are randomized into either of the groups to receive different modalities of post-operative PFMT.

Subjects in the S-PFMT group received traditional verbal instructions and paper-based educational materials. For the SI-PFMT group, an interactive experiential education model was adopted. First, an educational video introduced the importance and basic information of postoperative PFMT. Then, synchronized PFMT guidance through a combination of audio and video would be used. Subjects assigned to the S-PFMT+MS group, on the basis of traditional verbal and paper-based education, pelvic floor magnetic stimulation therapy was applied using a pelvic floor magnetic stimulator, operated by the same experienced rehabilitation physician.

Self administered questionnaires and 1-hour pad test would be used to assess the treatment outcomes at 1, 3, and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* PCa patients aged 18 to 85 years who had undergone laparoscopic radical prostatectomy (RP)

Exclusion Criteria:

* patients currently participating in other clinical trials and those unable to cooperate with study interventions and follow-up procedures due to specific factors

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | 1, 3, and 6 months postoperatively.
  A higher score indicates a more severe urinary incontinence and thus a worse outcome. Reduction in score is expected for subjects with clinical improvement.
  Range of score: 0 - 21 Severity of urinary incontinence: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21)

SECONDARY OUTCOMES:
urine leakage volume from the 1-hour pad test | 1, 3, and 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (2):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Arrangement not approved by national law of institute.